CLINICAL TRIAL: NCT03802513
Title: A New Therapeutic Approach for Somatosensory Tinnitus
Brief Title: Somatosensory Tinnitus Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3181-P; 1I21RX003181-01 (NIH)
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Tinnitus
Keywords: tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Individualized Physiotherapy (Other): This study has 1 health-related intervention. Veterans with somatosensory tinnitus will receive individualized physiotherapy.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Individualized physiotherapy including exercises to be performed by the Veteran at home.

SUMMARY:
Somatosensory tinnitus is suspected when the tinnitus perception changes following head, neck, or jaw maneuvers. The prevalence of this type of tinnitus in Veterans in unknown. The Cleveland Clinic evaluates all tinnitus patients for this condition and when detected, prescribes individualized physiotherapy. Cleveland Clinic's novel approach to tinnitus assessment and management provides the framework for this proof of concept pilot study.

DETAILED DESCRIPTION:
Phase 1A involves adapting Cleveland Clinic's assessment and treatment approach for somatosensory tinnitus to make it feasible for a VA population.

Phase 1B involves screening Veterans with tinnitus to evaluate and describe the prevalence of somatosensory tinnitus (in Veterans with tinnitus).

Phase 2 involves Veterans with somatosensory tinnitus receiving 3 individualized physical therapy sessions using the adapted approach developed during Phase 1A.

Phase 3 will evaluate the feasibility and tolerability of the adapted treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* chronic tinnitus
* positive screen for somatosensory tinnitus

Exclusion Criteria:

* Non-Veteran
* participation in new (< 1 month) tinnitus management or treatment
* current participation in tinnitus research involving an intervention

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Theodoroff, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individualized Physiotherapy
Started | 10
Completed | 9
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Individualized Physiotherapy
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Functional Index
Description: The TFI is a 25-item questionnaire that measures the functional effects of tinnitus. Total possible score ranges from 0-to-100 (scores >25 indicate tinnitus is a significant problem).
Time Frame: Baseline and 1 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individualized Physiotherapy
Number analyzed (Participants) | 9
score on a scale
  Baseline | 57.7 (22.3)
  1 month follow-up | 39.6 (26.0)

ADVERSE EVENTS:
Time Frame: The time frame for each participant's involvement in the study, and hence being monitored for adverse events, ranged from approximately 1 to 3 months.
Arm/Group | Individualized Physiotherapy
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
In-person research-related activities were limited due to COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03802513/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03802513/ICF_000.pdf